CLINICAL TRIAL: NCT00345189
Title: A Phase 1, Multicenter, Open-Label, Dose-Escalation, Safety, PK, and PD Study of CNF2024 Administered Orally Twice Weekly for 3 Weeks of a 4 Week Course or Twice Weekly for 4 Weeks of a 4 Week Course to Patients With Advanced Solid Tumors
Brief Title: Study of Oral CNF2024 (BIIB021) in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNF2024-ST-05003; 120ST101
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Tumors; Lymphoma
Keywords: Hsp90 inhibitor; CNF2024; Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — 6-chloro-9-(4-methoxy-3,5-dimethylpyridin-2-ylmethyl)-9H-purin-2-ylamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dosing Schedule 1 (Other): Starting dose of 25 mg, with dosing twice a week for 3 weeks out of a 4-week course (Schedule 1). Dosing for schedule 1 is currently closed.
  Interventions: Drug: CNF2024
- Dosing Schedule 2 (Other): Starting dose of 600 mg, with dosing twice a week for 4 weeks out of a 4-week course (without drug holidays; Schedule 2).
  Interventions: Drug: CNF2024

INTERVENTIONS:
Drug: CNF2024 — CNF2024 capsules administered orally following 2 schedules:
  * starting dose of 25 mg, twice a week for 3 weeks out of a 4-week course (Schedule 1) or
  * starting dose of 600 mg twice a week for 4 weeks out of a 4-week course (without drug holidays; Schedule 2).
  Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Dose escalation proceeds according to the predetermined scheme until the stopping dose is reached due to a dose limiting toxicity (DLT) occurring during the first 4-week course of treatment.
  Other Names: Advanced Solid Tumors

SUMMARY:
This is an open-label, multicenter, dose-escalation, safety, pharmacokinetics, and pharmacodynamics study.

DETAILED DESCRIPTION:
Heat shock protein 90 (Hsp90) is an ubiquitous molecular chaperone protein that is involved in folding, activation, and assembly of many proteins, including key mediators of signal transduction, cell cycle control, and transcriptional regulation. In cancer cells that are dependent upon Hsp90 client proteins, the degree to which clients are inhibited correlates closely with induction of growth inhibition and apoptosis with Hsp90 inhibitory drugs. The active pharmaceutical ingredient of CNF2024, CF1983 mesylate, is a synthetic, new chemical entity designed to inhibit Hsp90. CF1983 hada strong affinity for tumor derived Hsp90 and weaker affinity for Hsp90 isolated from normal cells or recombinant Hsp90.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor which has failed standard therapies (surgery, radiotherapy, endocrine therapy, chemotherapy) or for which effective therapy is not available
* At least 18 years of age
* Hematology: Absolute neutrophil count (ANC) > 1500 cells/mm3, platelet count > 100,000 cells/mm3 and hemoglobin >= 9 gm/L
* Hepatic: Bilirubin < 1.5 X upper limit of normal (ULN); alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5 X ULN. Patients with known liver metastases or liver neoplasms: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 5.0 X ULN.
* Renal: Serum creatinine levels < 2.0 mg/dL or creatinine clearance > 60 mL/min
* Coagulation: international normalized ratio (INR) < 1.5 times normal
* Adrenal: Normal plasma cortisol and adrenocorticotropic hormone (ACTH) levels
* Normal electrocardiogram (ECG) with QTc <= 450 msec for men and <= 470 msec for women
* Estimated life expectancy of at least 3 months as determined by the Investigator
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2
* Male and female patients of childbearing potential must practice effective double-barrier contraception during the study and continue contraception for 3 months after their last dose of study drug. Male patients must agree to not have intercourse with pregnant or nursing women during the study and for 3 months after their last dose of study drug, unless using double-barrier contraception. The only exceptions to double-barrier contraception are: Patient or partner is surgically sterile,female patient is postmenopausal for at least 1 year before screening or patient abstains from sexual intercourse, at the discretion of the Investigator

Exclusion Criteria:

* Pregnant or nursing women, women of child-bearing age not using reliable means of contraception.
* Radiotherapy or chemotherapy within the previous 28 days. Recovery to Grade 1 or less from chemotherapy-induced toxic effect, except alopecia, is required.
* Participation in any investigational drug study within 28 days prior to CNF2024 administration
* Active infection requiring intravenous antibiotic treatment
* Patients with second malignancy requiring active treatment (except hormonal therapy)
* Concurrent severe or uncontrolled medical disease (i.e., systemic infection, diabetes, hypertension, coronary artery disease, congestive heart failure)
* Active symptomatic fungal, bacterial and/or viral infection including active HIV or viral (A, B or C) hepatitis
* Problems with swallowing or malabsorption
* Chronic diarrhea (excess of 2-3 stools/day above normal frequency)
* Gastrointestinal diseases including gastritis, ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis
* Major surgery of the stomach or small intestine
* Adrenal dysfunction > Grade 2
* Patients with diabetes (your doctor will discuss if you are eligible for this study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-02; Primary Completion 2008-07 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) | Dose escalation will proceed according to the predetermined scheme until the stopping dose (dose > MTD) is reached due to dose limiting toxicities (DLT) occurring during the first 4-week course of treatment.
To determine the safety profile | Study duration
pharmacokinetic profile | Dosing period
effect on pharmacodynamic biomarkers | Dosing period
antitumor activity | At screening and after every 2 courses

CONTACTS AND LOCATIONS:
Overall Officials: Biogen Idec Medical Monitor, MD, Study Director — Biogen
Locations (4):
- United States (3):
  - Research site, Scottsdale, Arizona
  - Research site, New Haven, Connecticut
  - Research site, San Antonio, Texas
- Research site, Sutton, Surrey, United Kingdom